CLINICAL TRIAL: NCT02290548
Title: Effect of High-flow Nasal Oxygen vs Standard Oxygen Therapy on Extubation Outcome With High Risk of Extubation Failure in Medical ICU Patients
Brief Title: Effect of High-flow Nasal Oxygen on Extubation Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14MMHIS164
Record Dates: First submitted 2014-10-02; First posted 2014-11-14 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Failure; Congestive Heart Failure; COPD
Keywords: high flow nasal cannula; extubation failure
MeSH Terms: conditions — Respiratory Insufficiency; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high flow nasal cannula (Experimental): High flow nasal cannula immediately use after extubation
  Interventions: Device: high flow nasal cannula
- stanrd oxygen therapy (Placebo Comparator): Oxygen cannula or mask after extubation
  Interventions: Device: high flow nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula — High flow nasal cannula used in postextubation patients
  Other Names: Optiflow Airvo2 (Fisher & Paykel Healthcare)

SUMMARY:
The purpose of this study is to determine whether high flow nasal cannula is effective in lowering the reintubation rate after extubation for high risk patients in medical intensive care unit

DETAILED DESCRIPTION:
The study hypothesis is that Optiflow may reduce the extubation failure rate for high risk patients in medical intensive care unit.In the intervention group, patients fulfilling inclusion criteria and not presenting any of the exclusion criteria will receive high-flow nasal cannula (Optiflow Airvo2, Fisher & Paykel Healthcare Ltd., New Zealand) after extubation. The oxygen concentration (FiO2) will be set to reach an oxygenation target similar to control patients (see below), while the gas flow rate will be set at 50 L/min.In the control group, patients fulfilling inclusion criteria and not presenting any of the exclusion criteria will receive standard oxygen therapy including nasal cannula or oxygen mask after extubation. The FiO2 will be set to obtain a arterial oxygen saturation (SpO2) between 92% and 98% (or between 88% and 95% in hypercapnic patients). NIPPV or intubation will be applied in both group if respiratory distress noted. High flow nasal cannula will be tried before NIPPV or intubation in the control group patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients mechanically ventilated for > 48 hours and at least one of the following:
* > 65 y/o
* Cardiac failure as the primary indication of mechanical ventilation
* COPD
* Bronchiectasis
* Old pulmonary tuberculosis with destructive lung
* Chronic renal failure
* Neuromuscular disease
* BMI > 30
* Inability to manage respiratory secretions
* ARDS

Exclusion Criteria:

* Presence of tracheostomy
* Recent facial trauma
* Active gastro-intestinal bleeding
* Planned NIPPV support after extubation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
reintubation rate | 72 hours after extubation

SECONDARY OUTCOMES:
Need for Non-Invasive Ventilation | at day 28 after inclusion in the study
ICU readmission rate due to respiratory failure | at day 28 after inclusion in the study
ICU mortality rate | at day 28 after inclusion in the study
ICU length of stay | at day 28 after inclusion in the study
Hospital mortality | at day 28 after inclusion in the study
Hospital length of stay | at day 28 after inclusion in the study
Nosocomial pneumonia rate | at day 28 after inclusion in the study
Desaturation ( SaO2< 90%) | 72 hours after extubation
Severe hypoxemia (PaO2/Fraction of inspired O2 < 200) | Time Frame: 72 hours after extubation
hypercapnia (PaCO2 > 50) | 72 hours after extubation
respiratory acidosis (arterial pH < 7.30) | 72 hours after extubation
severe tachypnea (>40/min) | 72 hours after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Kuo Li Kuo, MD, Principal Investigator — +886975835135 lmn4093@gmail.com
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan